CLINICAL TRIAL: NCT05674175
Title: Use of Autologous Anti-CD22 CAR T Cells (CART22-65s) Co-administered With Humanized Anti-CD19 CAR T Cells (huCART19) in Children and Young Adults With Relapsed or Refractory B-ALL
Brief Title: Co-administration of CART22-65s and huCART19 for B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Chief, Cell Therapy and Transplant Section Director, Susan S. and Stephen P. Kelly Center for Cancer Immunotherapy Medical Director, Cell and Gene Therapy Lab, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-020640; 22CT015 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2022-12-06; First posted 2023-01-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B Lineage Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Finding Arm (Experimental): Phase 1 will evaluate the safety of co-administration of CART22-65s with huCART19 in patients who experienced a disease relapse after prior CAR T cell therapy. There is no planned dose escalation but a dose-deescalation will be made based on the incidence of Dose Limiting Toxicities
  Interventions: Biological: Autologous, humanized anti-CD22 CAR T cell therapy (CART22-65s); Biological: Autologous, humanized anti-CD19 CAR T cell therapy (huCART19)
- Expansion Arm (Experimental): If at least one dose level of phase 1 is determined to be safe, the phase 2 dose expansion phase of the trial will be opened to enrollment. Subjects will receive the highest dose of CART 22-65s and huCART19 cells that were determined to be safe. 2 cohorts are planned: Cohort A (relapsed/refractory, CAR T cell naïve) & Cohort B (prior treatment with a prior CAR T cell product).
  Interventions: Biological: Autologous, humanized anti-CD22 CAR T cell therapy (CART22-65s); Biological: Autologous, humanized anti-CD19 CAR T cell therapy (huCART19)

INTERVENTIONS:
Biological: Autologous, humanized anti-CD22 CAR T cell therapy (CART22-65s) — CART22-65s are autologous T cells that have been engineered to express an extracellular single chain antibody (scFv) with specificity for CD22 linked to an intracellular signaling molecule consisting of a tandem signaling domain comprised of the TCRζ signaling module linked to the 4-1BB costimulatory domain
  Other Names: CART22-65s
Biological: Autologous, humanized anti-CD19 CAR T cell therapy (huCART19) — HuCART19 cells are autologous T cells that have been engineered to express an extracellular single chain antibody (scFv) with specificity for CD19 linked to an intracellular signaling molecule consisting of a tandem signaling domain comprised of the TCRζ signaling module linked to the 4-1BB costimulatory domain
  Other Names: huCART19

SUMMARY:
This study will evaluate the safety and efficacy of administering two CAR T cell products, huCART19 and CART22-65s, in children with advanced B cell Acute Lymphoblastic Leukemia (B-ALL).

DETAILED DESCRIPTION:
CD19-targeted CAR T cell therapy has transformed the treatment landscape for children and young adults with chemo-refractory or relapsed B cell Acute Lymphoblastic Leukemia (B-ALL). Despite remarkable initial response rates, approximately 50% of pediatric patients experience a subsequent disease relapse. The prognosis for these patients is dismal with a median survival of less than one year from the time of post-CART19 relapse. The primary mechanisms contributing to CART19 failure include CD19-antigen escape and loss of CAR T cell surveillance due to short CART persistence. This study aims to counter each driver of relapse by co-administering two next-generation CAR T cell products: an anti-CD22 CART (CART22-65s), designed to overcome CD19-antigen escape; and a humanized anti-CD19 CART (huCART19), designed to overcome immune-mediated rejection of murine CART19.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Patients with documented CD19+ and/or CD22+ ALL/LLy:

   1. Cohort A: Patients with relapsed or refractory ALL/LLy:
   2. Cohort B: Patients with poor response to prior B cell directed engineered cell therapy
3. Patients with prior or current history of Central Nervous System 3 disease will be eligible if Central Nervous System disease is responsive to therapy
4. Documentation of CD19 and/or CD22 tumor expression in bone marrow, peripheral blood, Cerebrospinal fluid, or tumor tissue by flow cytometry at the time of last detectable disease. If the patient has experienced a relapse after CD19-directed and/or CD22-directed therapy, flow cytometry should be evaluated after this therapy to demonstrate CD19 and/or CD22 expression.
5. Age 0-29 years
6. Adequate organ function
7. Adequate performance status defined as Lanksy or Karnofsky performance score ≥50.
8. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria:

1. Active hepatitis B or active hepatitis C
2. HIV infection
3. Active acute or chronic Graft Vs. Host Disease requiring systemic therapy
4. Concurrent use of systemic steroids or immunosuppression at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy or immunosuppression during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
5. Central nervous system disease that is progressive on therapy, or with Central nervous system parenchymal lesions that might increase the risk of central nervous system toxicity.
6. Pregnant or nursing (lactating) women
7. Uncontrolled active infection

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Safety of CART22-65s and huCART19 co-administration | 1 year
  The safety of the administering CART22-65s and huCART19 will be measured by the monitoring the frequency and severity of adverse events in patients with advanced or refractory B-Cell Acute Lymphoblastic Leukemia or B Cell Lymphoblastic Lymphoma (B-LLy), including those previously treated with cell therapy.
Efficacy of CART22-65s and huCART19 co-administration | 1 year
  The efficacy of CART22-65s and huCART19 co-administration will be measured by the evaluating the overall response rate in patients with advanced or refractory B cell hematologic malignancies, including those previously treated with cell therapy.

SECONDARY OUTCOMES:
Manufacturing Feasibility | 5 years
  The manufacturing feasibility of manufacturing both CART22-65s and huCART19 will be measured by the percentage of manufactured products that do not meet release criteria for vector transduction efficiency, T cell product purity, viability, sterility or due to tumor contamination.
Anti-tumor response due to CART22-65s and huCART19 co-administration | Day 28
  Anti-tumor response due to CART22-65s and huCART19 co-administration will be measured by negative minimal residual disease (MRD) as measured by multiparameter flow cytometry at day 28.
Event Free Survival | 1 year
  1-year Event-Free Survival (EFS) in subjects with relapsed/refractory B-ALL (Cohort A) and in subjects with poor response to prior B cell directed engineered cell therapy (Cohort B)
Relapse Free Survival | 1 year
  1-year relapse-free survival (RFS) rate in CAR-naïve subjects with relapsed/refractory B-ALL (Cohort A) and in CAR-exposed subjects with poor response to prior B cell directed engineered cell therapy (Cohort B)
Overall Survival | 1 year
  1-year overall survival (OS) rate in CAR-naïve subjects with relapsed/refractory B-ALL (Cohort A) and in CAR-exposed subjects with poor response to prior B cell directed engineered cell therapy (Cohort B).
CAR T Cell Therapy Persistence | 1 year
  CART22-65s and huCART19 persistence polymerase chain reaction (or flow cytometry) analysis of whole blood to detect and quantify survival of CART2265s and huCART19 over time.
Bioreactivity of CART22-65s and huCART19 when co-administered | 1 year
  The bioreactivity of CART22-65s and huCART19 when co-administered, as measured by elevations level in any of; Uric Acid, Lactate Dehydrogenase (LDH), c-reactive protein (CRP), and cytokines (e.g.IL -10) before and after CART T cell infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Myers, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No